CLINICAL TRIAL: NCT00779727
Title: Post-Cesarean Wound Drainage is Not Necessary in Women at Increased Risk of Hemorrhage
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05/99
Record Dates: First submitted 2008-09-04; First posted 2008-10-24 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2008-09

CONDITIONS: Pregnancy; Hemorrhage
Keywords: women; increased; risk
MeSH Terms: conditions — Hemorrhage

INTERVENTIONS:
Procedure: Placement of drainages

SUMMARY:
Randomized controlled trial assessing the benefit of cesarean wound drainage in pregnant women at increased risk of hemorrhage. The pregnant women at increased risk of hemorrhage were randomised in two groups. In one group 2 wound drainages were placed during the cesarean section, in the other group none. Outcome measures were difference between preoperative and postoperative hemoglobin, postoperative fever, cumulative opiate dose adjusted to body weight, length of stay and operation time. It is postulated that the pregnant women with increased risk of hemorrhage do not profit from the routine placement of wound drainages.

* Trial with surgical intervention

ELIGIBILITY:
Inclusion criteria:

* All pregnant women with increased risk of hemorrhage carrying singleton pregnancies, who had to undergo cesarean section.

Exclusion criteria:

* Twin-pregnancies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-10; Study Completion 2004-06

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland